CLINICAL TRIAL: NCT00203827
Title: Pediatric Sleep Questionnaire: Use for Collection of Clinical Data
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13272A
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep Disorders
Keywords: Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a questionnaire that can be used for standardized patient information gathering in the clinical setting. This will serve as the information source for a pediatric sleep database.

DETAILED DESCRIPTION:
A sleep questionnaire will be administered to patients who present to the Pediatric Neurology Clinic and the Pediatric Sleep Clinic in the DCAM as well as LaRabida Children's Hospital complaining of sleep problems. The questions asked are those routinely obtained in clinical practice of sleep medicine. Medical students, residents and faculty as part of their normal clinical responsibilities will administer the questionnaire. The database will be maintained in Filemaker Pro program for future research purposes. Collection of the data will require approximately 15 minutes. A database file number not related to the patient medical record number will be assigned to each patient. The investigator will keep a separate log linking patient database number and patient medical record number. The logbook will be kept under lock and key by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen in the Pediatric Neurology Clinic and at La Rabida Children's Hospital

Exclusion Criteria:

* Adults

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Problems or habits children experience with sleep
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pediatric Sleep Questionnaire | When data from clinic patients becomes available
  This questionnaire is used to better understand the natural history of sleeping disorders in children.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kohrman, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States